CLINICAL TRIAL: NCT04652700
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate the Efficacy and Safety of Oral Islatravir Once-Monthly as Preexposure Prophylaxis in Cisgender Men and Transgender Women Who Have Sex With Men, and Are at High Risk for HIV-1 Infection
Brief Title: Oral Islatravir (MK-8591) Once-Monthly as Preexposure Prophylaxis (PrEP) in Men and Transgender Women Who Are at High Risk for HIV-1 Infection (MK-8591-024)
Acronym: Impower-024
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Voluntarily terminated due to benefit/risk assessment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8591-024; MK-8591-024 (Other: MSD); jRCT2031200419 (Registry Identifier: jRCT); 2020-003309-79 (EudraCT Number)
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: HIV Preexposure Prophylaxis
Keywords: Preexposure prophylaxis (PrEP); Prevention
MeSH Terms: interventions — islatravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In Study Part 1, double-blind with in-house blinding is used.
  In Study Part 2, sponsor personnel not directly involved with blinded safety monitoring will be unblinded to participants' randomized study intervention in Part 1 (personnel involved with Part 2 will remain blinded).
  In Study Part 3, al participants, investigators, and Sponsor personnel are unblinded as to the participant's original randomized intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Islatravir (ISL) Once Monthly (QM) Group (Experimental): Participants receive 60 mg tablet of ISL QM, orally plus Placebo to Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) tablet once daily (QD) or Placebo to Emtricitabine/Tenofovir Alafenamide (FTC/TAF) tablet QD, orally for up to 24 months of treatment duration.
  Interventions: Drug: ISL; Drug: Placebo to FTC/TDF; Drug: Placebo to FTC/TAF
- FTC/TDF or FTC/TAF QD Group (Active Comparator): Participants receive 200/245 mg or 200/300 mg of FTC/TDF combination tablet, QD, orally or 200/25 mg of FTC/TAF combination tablet, QD, orally at investigator's discretion plus Placebo to ISL tablet QM, orally for up to 24 months of treatment duration.
  Interventions: Drug: FTC/TDF; Drug: FTC/TAF; Drug: Placebo to ISL

INTERVENTIONS:
Drug: ISL — ISL 60 mg tablet, QM, orally for up to 24 months
  Other Names: MK-8591
  Arms: Islatravir (ISL) Once Monthly (QM) Group
Drug: FTC/TDF — Participants receive 200/245 mg of FTC/TDF combination tablet, QD, orally for up to 24 months
  Other Names: Truvada; Emtricitabine/Tenofovir Disoproxil Fumarate
  Arms: FTC/TDF or FTC/TAF QD Group
Drug: FTC/TAF — Participants receive 200/25 mg of FTC/TAF combination tablet, QD, orally for up to 24 months
  Other Names: Descovy; Emtricitabine/Tenofovir Alafenamide
  Arms: FTC/TDF or FTC/TAF QD Group
Drug: Placebo to ISL — Placebo ISL 0 mg tablets QM, orally for up to 24 months.
  Arms: FTC/TDF or FTC/TAF QD Group
Drug: Placebo to FTC/TDF — Placebo FTC/TDF 0 mg tablets QD, orally for up to 24 months
  Arms: Islatravir (ISL) Once Monthly (QM) Group
Drug: Placebo to FTC/TAF — Placebo FTC/TAF 0 mg tablets QD, orally for up to 24 months
  Arms: Islatravir (ISL) Once Monthly (QM) Group

SUMMARY:
The main purpose of the study is to evaluate the safety and tolerability of oral Islatravir (ISL) once monthly (QM) as Preexposure Prophylaxis (PrEP) in cisgender men who have sex with men (MSM) and transgender women (TGW) who have sex with men and who are at high risk of HIV-1 infection with 48 or 96 weeks of treatment and a minimum follow-up of 42 days.

DETAILED DESCRIPTION:
Based on laboratory findings of decreased lymphocyte and CD4+ T-cell counts across the islatravir program, dosing of blinded study intervention was halted on 13-Dec-2021. Blinded assessments conducted prior to then are designated as Study Part 1. During Study Part 2, participants from Part 1 were switched to PrEP therapy with emtricitabine/tenofovir disoproxil (FTC/TDF) or emtricitabine/tenofovir alafenamide (FTC/TAF) while continuing in the study, but participants, investigators, and Sponsor personnel remained blinded to the Part 1 treatment. In Part 3, participants, investigators, and all Sponsor personnel are unblinded to participant's original randomized intervention group, and participants may continue to receive unblinded FTC/TDF or FTC/TAF.

ELIGIBILITY:
Inclusion Criteria:

* Has confirmed Human Immunodeficiency Virus (HIV) uninfected based on negative HIV-1/HIV-2 test result before randomization
* Is sexually active with male or transgender women (TGW) partners defined as having anal sexual intercourse with a man or TGW at least once in the past month
* Is at high risk for sexually acquiring HIV-1 infection based on self-report of at least 1 of the following: a) Condomless receptive anal intercourse in the 6 months prior to screening occurring outside a mutually monogamous HIV seronegative concordant relationship b) More than 5 partners (anal intercourse) in the 6 months prior to screening c) Any unprescribed stimulant drug use in the 6 months prior to screening d) Rectal or urethral gonorrhea or chlamydia or incident syphilis in the 6 months prior to screening
* Participants 16 or 17 years of age must weigh ≥35 kg. Enrollment for 16- to 17-year-old participants will begin only after completion of the Sentinel Cohort IA and review of IA results by the external data monitoring committee (eDMC)
* Has no plans to relocate or travel away from the site for ≥4 consecutive weeks during study participation

Exclusion Criteria:

* Has hypersensitivity or other contraindication to any component of the study interventions as determined by the investigator
* Has chronic HBV infection or past HBV infection which could indicate risk for Hepatitis B reactivation
* Has known current or chronic history of liver disease or known hepatic or biliary abnormalities, unless the participant has stable liver function tests and no evidence of hepatic synthetic dysfunction
* Has a history of malignancy within 5 years of screening except for adequately treated basal cell or squamous cell skin cancer or in situ anal cancers
* Has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might, in the opinion of the investigator, confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to enroll
* Has taken cabotegravir, lenacapavir, or any other long-acting HIV prevention product at any time
* Is currently receiving or is anticipated to require any prohibited therapies outlined in the study from 30 days prior to Day 1 through the duration of the study
* Is currently participating in or has participated in an interventional or prevention clinical study with an investigational compound or device, within 30 days prior to Day 1 through the duration of the study
* Has exclusionary laboratory values within 45 days prior to Day 1

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants and transgender women (TGW) who are at high risk for HIV-1 infection
Enrollment: 494 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- United States (15):
  - University of Alabama at Birmingham-UAB 1917 Research Clinic ( Site 0007), Birmingham, Alabama
  - UCLA Center for Clinical AIDS Research and Education ( Site 0011), Los Angeles, California
  - Global Research Institute ( Site 0031), Los Angeles, California
  - Bridge HIV - San Francisco Department of Public Health ( Site 0003), San Francisco, California
  - The GW Medical Faculty Associates-Medicine ( Site 0033), Washington D.C., District of Columbia
  - Midway Immunology and Research Center ( Site 0014), Ft. Pierce, Florida
  - University of Miami Miller School of Medicine-Infectious Disease ( Site 0029), Miami, Florida
  - Orlando Immunology Center ( Site 0010), Orlando, Florida
  - Ponce De Leon Center Grady Health ( Site 0032), Atlanta, Georgia
  - Howard Brown Health Center ( Site 0004), Chicago, Illinois
  - The University of Mississippi Medical Center ( Site 0012), Jackson, Mississippi
  - Rutgers New Jersey Medical School-Clinical Research Center ( Site 0017), Newark, New Jersey
  - The University of North Carolina at Chapel Hill ( Site 0019), Chapel Hill, North Carolina
  - Central Texas Clinical Research ( Site 0002), Austin, Texas
  - The Crofoot Research Center ( Site 0025), Houston, Texas
- Centro de Referência e Treinamento DST/AIDS ( Site 0351), São Paulo, Brazil
- Hôpital Saint-Louis-Infectious Diseases and tropical diseases ( Site 0151), Paris, Île-de-France Region, France
- Center Hospital of the National Center for Global Health and Medicine ( Site 0101), Shinjyuku-ku, Tokyo, Japan
- Via Libre ( Site 0404), Lima, Peru
- South Africa (3):
  - Perinatal HIV Research Unit (PHRU)-HIV Prevention CRS ( Site 0203), Johannesburg, Gauteng
  - Wits Reproductive Health and HIV Institute (WRHI)-Research Center ( Site 0201), Johannesburg, Gauteng
  - Desmond Tutu HIV Foundation ( Site 0202), Cape Town, Western Cape
- Thailand (3):
  - Chulalongkorn University-Pediatrics ( Site 0051), Bangkok, Bangkok
  - HIV Netherlands Australia Thailand Research Collaboration ( Site 0056), Bangkok, Bangkok
  - Research Institute for Health Sciences-Research Institute for Health Sciences Building 1 ( Site 0052, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26375&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized at 23 study sites in France, Japan, Peru, South Africa, and the United States.
Groups:
- Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF: Participants received 60 mg tablet of ISL once monthly (QM) plus placebo to FTC/TDF tablet once daily (QD) or placebo to FTC/TAF tablet QD in Part 1. Participants then received open-label FTC/TDF or FTC/TAF in Parts 2 and 3.
- Parts 1 to 3: FTC/TDF or FTC/TAF: Participants received 200/245 mg or 200/300 mg of FTC/TDF combination tablet QD or 200/25 mg of FTC/TAF combination tablet QD at investigator's discretion plus placebo to ISL tablet QM in Part 1. Participants continued to receive open-label FTC/TDF or FTC/TAF in Parts 2 and 3.
Period: Part 1: Blinded Study Medication
Arm/Group | Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF | Parts 1 to 3: FTC/TDF or FTC/TAF
Started (Started randomized treatment) | 328 | 166
Completed | 0 | 0
Not Completed | 328 | 166
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 7 | 2
Not completed — Multiple reasons (primarily discontinuation of blinded treatment) | 308 | 160
Not completed — Withdrawal by Subject | 12 | 4
Period: Parts 2 and 3: Open-Label FTC TDF or TAF
Arm/Group | Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF | Parts 1 to 3: FTC/TDF or FTC/TAF
Started (Started optional open-label therapy) | 306 | 154
Completed | 0 | 0
Not Completed | 306 | 154
Not completed — Lost to Follow-up | 34 | 9
Not completed — Not reported | 6 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Study terminated by Sponsor | 227 | 119
Not completed — Withdrawal by Subject | 39 | 23

BASELINE CHARACTERISTICS:
Groups:
- Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF: Participants received 60 mg tablet of ISL QM plus placebo to FTC/TDF tablet QD or placebo to FTC/TAF tablet QD in Part 1. Participants then received open-label FTC/TDF or FTC/TAF in Parts 2 and 3.
- Total: Total of all reporting groups
Arm/Group | Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF | Parts 1 to 3: FTC/TDF or FTC/TAF | Total
Number analyzed (Participants) | 328 | 166 | 494
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (9.6) | 29.5 (9.2) | 29.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 328 | 166 | 494
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 111 | 51 | 162
  Not Hispanic or Latino | 214 | 111 | 325
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 70 | 31 | 101
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 83 | 41 | 124
  White | 135 | 71 | 206
  More than one race | 35 | 20 | 55
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE) During Blinded Treatment
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced an AE will be reported for each treatment arm.
Time Frame: Up to approximately 10.5 months
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF | Parts 1 to 3: FTC/TDF or FTC/TAF
Number analyzed (Participants) | 328 | 166
Participants | 211 | 128

2. Primary Outcome: Number of Participants Who Discontinued From Blinded Study Treatment Due to an AE
Description: as for outcome 1
Time Frame: Up to approximately 9 months
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF | Parts 1 to 3: FTC/TDF or FTC/TAF
Number analyzed (Participants) | 328 | 166
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Confirmed HIV-1 Infection
Description: The number of participants with confirmed HIV-1 infections during the blinded treatment period is presented.
Time Frame: Up to approximately 10.5 months
Population: All participants who were randomized and received ≥1 dose of study intervention are included (participants with confirmed HIV infections prior to or at randomization are excluded).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: ISL & Parts 2 & 3: FTC/TDF or FTC/TAF | Parts 1 to 3: FTC/TDF or FTC/TAF
Number analyzed (Participants) | 328 | 166
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Entire Study: Blinded Treatment (Part 1) + Open-Label Standard-of-Care Treatment (Parts 2 & 3) [Up to approximately 26 months]
Description: All treated participants are included. Data are presented separately for Part 1 (randomized blinded treatment) and Parts 2 & 3 (open-label standard-of-care preexposure prophylaxis [PrEP] periods). Open-label PrEP treatment was pooled per protocol as standard-of-care treatment (FTC/TAF as available only for US sites, FTC/TDF as brand [200/300 mg] or generic [200/245 mg]).
Groups:
- Part 1: ISL: Participants received blinded 60 mg tablet of ISL QM plus placebo to FTC/TDF tablet QD or placebo to FTC/TAF tablet QD in Part 1.
- Parts 2 & 3: Open-label PrEP (ISL in Part 1): Participants received open-label FTC/TDF or FTC/TAF (based on regional availability) QD in Parts 2 and 3 (after blinded ISL in Part 1).
- Part 1: FTC/TDF or FTC/TAF: Participants received blinded FTC/TDF (200/245 mg or 200/300 mg) or FTC/TAF (200/25 mg) QD in Part 1.
- Parts 2 & 3: Open-label PrEP (FTC/TDF or FTC/TAF in Part 1): Participants received open-label FTC/TDF or FTC/TAF (based on regional availability) QD in Parts 2 and 3 (after blinded FTC/TDF or FTC/TAF in Part 1).
Arm/Group | Part 1: ISL | Parts 2 & 3: Open-label PrEP (ISL in Part 1) | Part 1: FTC/TDF or FTC/TAF | Parts 2 & 3: Open-label PrEP (FTC/TDF or FTC/TAF in Part 1)
All-Cause Mortality (participants affected / at risk) | 0/328 | 0/306 | 0/166 | 0/154
Serious Adverse Events (participants affected / at risk) | 6/328 | 18/306 | 1/166 | 5/154
Other Adverse Events (participants affected / at risk) | 120/328 | 230/306 | 88/166 | 104/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ISL (N=328) | Parts 2 & 3: Open-label PrEP (ISL in Part 1) (N=306) | Part 1: FTC/TDF or FTC/TAF (N=166) | Parts 2 & 3: Open-label PrEP (FTC/TDF or FTC/TAF in Part 1) (N=154)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 8 (8) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ISL (N=328) | Parts 2 & 3: Open-label PrEP (ISL in Part 1) (N=306) | Part 1: FTC/TDF or FTC/TAF (N=166) | Parts 2 & 3: Open-label PrEP (FTC/TDF or FTC/TAF in Part 1) (N=154)
Diarrhoea (Gastrointestinal disorders) | 19 (21) | 14 (14) | 9 (11) | 11 (11)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 12 (12) | 2 (2) | 8 (9)
COVID-19 (Infections and infestations) | 35 (36) | 69 (79) | 21 (21) | 37 (41)
Chlamydial infection (Infections and infestations) | 0 (0) | 17 (19) | 2 (2) | 7 (9)
Influenza (Infections and infestations) | 4 (4) | 14 (19) | 6 (7) | 14 (15)
Latent syphilis (Infections and infestations) | 2 (2) | 18 (22) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 14 (14) | 27 (33) | 7 (8) | 11 (12)
Oropharyngeal gonococcal infection (Infections and infestations) | 16 (18) | 41 (55) | 11 (11) | 24 (29)
Pharyngeal chlamydia infection (Infections and infestations) | 2 (2) | 18 (18) | 1 (1) | 2 (2)
Proctitis chlamydial (Infections and infestations) | 20 (25) | 65 (81) | 14 (14) | 27 (37)
Proctitis gonococcal (Infections and infestations) | 13 (14) | 51 (63) | 15 (16) | 30 (41)
Syphilis (Infections and infestations) | 10 (10) | 19 (20) | 7 (7) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 31 (32) | 8 (8) | 17 (20)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 24 (29) | 3 (3) | 6 (10)
Headache (Nervous system disorders) | 14 (14) | 18 (23) | 10 (10) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 16 (17) | 3 (3) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (15) | 7 (8) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT04652700/Prot_SAP_000.pdf